CLINICAL TRIAL: NCT01011127
Title: Different Metabolic Effects of Statins
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Other Study IDs: GMC-200914
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Hypercholesterolemia
Keywords: Statins; Insulin resistance
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pravastatin
  Interventions: Drug: pravastatin, rosuvastatin
- rosuvastatin
  Interventions: Drug: pravastatin, rosuvastatin

INTERVENTIONS:
Drug: pravastatin, rosuvastatin

SUMMARY:
The investigators hypothesize that pravastatin and rosuvastatin may have different metabolic effects in hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein cholesterol levels>130

Exclusion Criteria:

* Overt liver disease Chronic renal failure Hypothyroidism Myopathy Uncontrolled diabetes Severe hypertension

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hypercholesterolemia
Sampling Method: Probability Sample
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Background] Yada T, Nakata M, Shiraishi T, Kakei M. Inhibition by simvastatin, but not pravastatin, of glucose-induced cytosolic Ca2+ signalling and insulin secretion due to blockade of L-type Ca2+ channels in rat islet beta-cells. Br J Pharmacol. 1999 Mar;126(5):1205-13. doi: 10.1038/sj.bjp.0702397. PMID 10205010